CLINICAL TRIAL: NCT01005498
Title: Comparison Between Low Carbohydrate Diet and Traditionally Recommended Diabetic Diet in the Treatment of Diabetes Mellitus Type 2.
Acronym: VÄSTKOST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vårdcentralen Lyckorna (Other)
Responsible Party: Principal Investigator, Hans Guldbrand, Distriktsläkare, Vårdcentralen Lyckorna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M216-08
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes
Keywords: Low carbohydrate diet. Dietary treatment of diabetes mellitus.; Diabetes mellitus type 2 and dietary treatment.
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low carbohydrate diet (F) (Experimental): The group attended to low carbohydrate diet
  Interventions: Dietary Supplement: Low carbohydrate - high fat diet
- Traditional diet (K) (Active Comparator): The group attended to traditional diet
  Interventions: Dietary Supplement: High carbohydrate - low fat diet

INTERVENTIONS:
Dietary Supplement: Low carbohydrate - high fat diet — The diet has an energy content of 1600 kcal or 1800, with 50% from fat, 20% from carbohydrates and 30% from proteins.
  Arms: Low carbohydrate diet (F)
Dietary Supplement: High carbohydrate - low fat diet — The diet has an energy content of 1600 or 1800 kcal, with 30% from fat, 55-60% from carbohydrates and 10-15% from proteins.
  Arms: Traditional diet (K)

SUMMARY:
The purpose of the clinical trial is to investigate whether low carbohydrate diet is better than the traditional diabetic diet in the treatment of patients with diabetes mellitus type 2, for blood sugar and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2

Exclusion Criteria:

* Severe psychiatric disease or difficulties in understanding Swedish language.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Laboratory findings and body composition | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans G Guldbrand, Principal Investigator — Vårdcentralen Lyckorna
Locations (1):
- Vårdcentralen Lyckorna, Motala, Östergötland County, Sweden

REFERENCES:
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 Aug 21;8(8):CD011737. doi: 10.1002/14651858.CD011737.pub3. PMID 32827219
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 May 19;5(5):CD011737. doi: 10.1002/14651858.CD011737.pub2. PMID 32428300
- [Derived] Guldbrand H, Dizdar B, Bunjaku B, Lindstrom T, Bachrach-Lindstrom M, Fredrikson M, Ostgren CJ, Nystrom FH. In type 2 diabetes, randomisation to advice to follow a low-carbohydrate diet transiently improves glycaemic control compared with advice to follow a low-fat diet producing a similar weight loss. Diabetologia. 2012 Aug;55(8):2118-27. doi: 10.1007/s00125-012-2567-4. Epub 2012 May 6. PMID 22562179